CLINICAL TRIAL: NCT05429619
Title: Advancing Peer Support Programming to Address PTSD and Trauma Among Canadian Public Safety Personnel and Veterans
Brief Title: Evaluating Implementation and Impact of PeerOnCall, a Mobile Health Approach to Peer Support for Canadian Public Safety Personnel
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: University of Regina (Other); Canadian Institute for Public Safety Research and Treatment (Unknown); Public Health Agency of Canada (PHAC) (Other Government); Wilfrid Laurier University (Other); Memorial University of Newfoundland (Other); Western University (Other); Fisheries and Marine Institute of Memorial University of Newfoundland (Unknown)
Responsible Party: Sponsor
Other Study IDs: 14731
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Issue; Mental Stress; Post Traumatic Stress Disorder
Keywords: peer support; mobile health
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PeerOnCall — A mobile health peer-to-peer support platform that consists of two inter-connected apps: PeerOnCall and PeerOnCall Support. The apps were co-designed by and for the public safety community in Canada, with customized content for correctional workers, emergency communicators, firefighters, paramedics and police.
  Other Names: PeerOnCall Support

SUMMARY:
A prospective cohort study design will be implemented across four sectors and multiple organizations sites to evaluate implementation and impact of the apps. Pre/post impact data will be collected over a six-month implementation period to assess whether the apps lead to increased Public Safety Personnel outreach to peer support (primary outcome), and to increased mental health literacy, and decreased mental distress (secondary outcomes). Recruitment will take place at three levels; 1) organizations (including knowledge users/organization champions), 2) peer support providers, and 3) public safety personnel employed within each participating organization. Sources of implementation and impact data for the six-month trial will include: 1) app utilization data, 2) knowledge user/organization champion interviews, 3) surveys with public safety personnel, 4) focus groups with peer support providers, and 5) implementation costs. Analysis will focus on both implementation and effectiveness to address the research questions related to the impact of the apps, as well as how the process and context of implementation shapes effectiveness.

DETAILED DESCRIPTION:
PeerOnCall was developed to support frontline PSP and includes features such as anonymous calling or messaging to a choice of peer support providers, access to self-screening tools, a personal wellness toolbox, and "tips to cope" resources. PeerOnCall Support is designed for peer support providers to provide a secure, private platform for providing support to peers who reach out via text or telephone through the PeerOnCall app.

This study will explicitly scale implementation and evaluation of these apps in the context of day-to-day work within a range of PSP organizations across four different service sectors (corrections, emergency communicators, fire services and paramedic services).

The implementation period for the app is six-months. Prior to the end of the six-month implementation period, the sector lead will meet with each organization to review app utilization data and to discuss options for continued usage of the app within the organization.

The Consolidated Framework for Implementation Research (CFIR) will inform exploration, not only of whether the apps 'work', but also about how the apps are adopted, and the individual and organizational forces that shape adoption.

The study will deploy the apps to a purposive sample of approximately 24 organizations across four sectors: 1) correctional workers; 2) emergency communicators (e.g., 911 call takers, dispatchers); 3) fire services; and 4) paramedic services. All participating organizations must have an established internal peer support service (with procedures for vetting, training, and ongoing support of the peer support providers), an organization champion who will liaise between the research team and employees, and support from leadership to participate in the study. The process of recruitment will be facilitated by sector leads and knowledge users who have extensive networks within the sectors. The number of organizations recruited across each sector will be different, recognizing differences in how services are provided, and the need for understanding breadth versus depth of implementation in key stakeholder groups.

Within each sector, key knowledge users (at the sector level) and organization champions (at the organization level) will be recruited. The sector-level knowledge users will provide insights into general considerations for implementation and evaluation. In the participating organizations, one or two "champions" will be recruited who will be responsible for organization onboarding, including customizing content, securing participation of in-house peer support providers, and sharing information with co-workers via formal and informal communication channels.

Peer support providers within each organization will be recruited to provide services through the app. All trained peer providers within each organization will be invited to participate. Information meetings will be held in each organization for the peer supporters regarding the PeerOnCall Support app. The orientation will ensure that the peer supporteres are aware of how to use the app and the protocols for responding to PSP who reach out for support, including those who may be in crisis.

All eligible employees within each organization will be invited to participate in the research via established communication channels within the organization (e.g., recruitment posters distributed via email, social media etc.), and information meetings held in the organization in the month prior to distributing access to the PeerOnCall app. After orientation within the organization, employees will be provided with an organization code to access the PeerOnCall app once it has been downloaded from the Google Play or Apple store. Employees can choose whether to download the app and they are able to use the app without engaging in the baseline and follow-up surveys.

To ensure adequate power for evaluating impact of the app, sample size estimates were based on the primary outcome of interest: the frequency of outreach to peer support through the app (count of the number of times contact was initiated by PeerOnCall users via phone and/or text). The sample size was calculated using a one-sided Poisson test since the frequency of outreach via the app can only increase from no outreach at baseline. Assuming 90% power, a significance level of 0.025 for a one-sided test, a hypothesized rate of 0.2 (20% increase in rates of outreach) and alternative hypothesis rate of 0.1 (thus a difference of 0.1), 161 participants will be required. Considering an estimated 20% drop out rate, 202 participants will be needed.

Aggregate data collected will include participant adoptions rates across each organization (e.g., the number of times the app was downloaded) as well as aggregate data on how often the app was used, average durations of use, the number of times different features were accessed, and the number and duration of contacts with peer supporters.

Knowledge user/Organization Champion Interviews will be conducted at baseline, three-months and six-months after app implementation begins at each participating organization to explore the context for implementation. Interview questions will be congruent with the Consolidated Framework for Implementation Research. These data will be used to identify facilitators and barriers to app use and inform interpretation of the adoption rates and outcome data both within and across participating organizations.

To track immediate feedback about the peer support service, a 'pop-up' feedback survey is presented to users within the application following each peer support encounter asking for a rating of their level of distress before and after the interaction using a 10-point Visual Analogue Scale. There is also an option to provide comments about the encounter. Data from the feedback surveys will help understand the immediate impact of peer support on level of distress.

To evaluate user impact over time, employees in each organization will be invited to complete baseline, three-month, and six-month follow-up surveys via a link to complete a survey.

Focus groups will be scheduled at three-months and six months after the implementation period with PeerOnCall Support peer support providers to explore their experiences with providing peer support through the app. Three sets of focus groups will be conducted within each sector with six to eight participants in each group.

Data regarding implementation costs within each organization will include: the organization champion's time invested on onboarding and communication, administrative time for uploading users and responding to requests, and metrics regarding peer support service provision. The cost of server hosting, troubleshooting, and regular upgrades to the apps will also be tracked across sites.

Implementation within each organization will be tracked via descriptive data regarding adoption rates (proportion of employees who download & use the app), and usage rates over time, including the number of times users reach out for peer support via phone/text, and the number of repeated calls.

To evaluate effectiveness, analysis of the pre/post survey data will examine the change in scores across the dataset in dimensions of mental health literacy, levels of mental distress (standardized assessments of anxiety, depression, and Post Traumatic Stress Disorder), and frequency of outreach behaviors in seeking mental health support. Multiple hierarchical linear regression analyses will be conducted to examine differences in effectiveness based on gender, service, and job tenure.

Effectiveness of the peer support service will also be evaluated by comparing change scores in level of distress before and after each peer support encounter via the in-app surveys.

Identification of barriers and facilitators to adoption of the technology and peer support service will occur through qualitative content analysis of the interview transcripts with the organizational champions and focus groups with the peer supporters. The CFIR framework will guide the analysis process considering organization internal and external forces, as well as how communication strategies influence implementation, and consistency in providing the peer support service.

All the data from the evaluation process will be reviewed to generate recommendations for optimizing uptake and impact of the app across different types of organizations.

ELIGIBILITY:
Inclusion Criteria:

* Public Safety Personnel working in fire services, paramedic services, emergency communications and correctional services
* Employed (full or part-time) by the participating organizations
* Agree to download the PeerOnCall app on their mobile phone (Android or Apple)

Exclusion Criteria:

- Not able to access the app on their mobile health device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals employed by participating Public Safety Organizations (fire services, paramedic services, emergency communications, correctional services).
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Accessing peer support via phone or text via the PeerOnCall app (Frequency count) | Monthly intervals from 1 to 6 months.
  Number of times PeerOnCall users within an organization create a connection with peer support providers via the app platform (Software analytics)

SECONDARY OUTCOMES:
Change in Mental Health Literacy (6 items, 7-point Likert scale rating) | Baseline, 3 months, 6 months
  Rating using a 7-point Likert scale of perceived improvement in dimensions of mental health literacy (Promote mental health, knowledge of how to identify and address mental health issues in self and others, how to identify relevant resources). Range 7-42 with higher scores indicating higher levels of perceived literacy.
Changes in symptoms of anxiety (GAD-7 screening tool) | Baseline, 3 months, 6 months
  The Generalised Anxiety Disorder (GAD-7) scale is a 7-item tool to evaluate anxiety symptoms over the past two weeks (4-point Likert scale ratings). Scores ranges from 0-21 with a score of 10 or more indicative of potential generalized anxiety disorder.
Change in symptoms of depression (PHQ-9 screening tool) | Baseline, 3 months, 6 months
  The Patient Health Questionnaire (PHQ-9) is a 9-item screening tool for depression. Scores range from 0-27, with a score of 10 or more indicative of major depression.
Change in symptoms of trauma (PTSD Checklist, PCL-5 short version) | Baseline, 3 months, 6 months
  The short version of the Post-Traumatic Stress Disorder Checklist (PCL-5) is a four-item PTSD screening checklist exploring responses to a stressful experience in terms of symptoms over the past month. Scores range from 0-16 with higher scores indicating more severe impairment.
Change in help-seeking behaviour | Baseline, 3 months, 6 months
  Rating of how likely to reach out for support related to four different types of support (In-person peer support, app-based peer support, professional support, and employee assistance program). Ratings on a 5-point scale from not at all likely to extremely likely.
Perceived value of the app | 3 months, 6 months
  Questions about perceived impact adapted from the Mobile Rating Application Rating Scale (MARS) asks users to rate (on a 5-point Likert scale) the perceived value of the app on 7 items (Awareness of the importance of addressing mental health, reaching out for help and impact on mental health, perceived support, and ability to cope at work).
Change in perceived level of stress | Baseline, 3 months, 6 months
  Rating of current level of stress on a 7-point Likert scale from very low to very high.
Change in perceptions of workplace psychological health and safety climate | Baseline, 3 months, 6 months
  Rating of psychological health and safety climate in the workplace on a 7-point Likert scale from toxic to excellent.
Change in current mental health challenges | Baseline, 3 months, 6 months
  Rating of current mental health challenges on a 100-point Visual Analogue scale from ill to healthy.
Impact on work | Baseline, 3 months, 6 months
  Questions about the number of hours users were scheduled/expected to work and the number of hours of work users missed because of the way they were feeling over the past 2 weeks.

OTHER OUTCOMES:
Digital literacy | Baseline, 3 months, 6 months
  Rating of knowledge and comfort level in using apps. Ratings from low to high levels of digital literacy. Hypothesis is that lower digital literacy will predict lower app use. The baseline scale provides descriptive data about levels of digital literacy across the organization. The follow-up scale provides descriptive data about perceived digital literacy.
Frequency of app use | 3 months, 6 months
  Report of how often the app was used over the past 4 weeks, ranging from not at all to more than once a day. This data can be used to note dose/response (I.e., Higher app use might lead to greater impact) and to track app user over time.
Timing of app use | 3 months, 6 months
  Descriptive data of when the app is used the most. Can be used to report trends within/across sectors and organizations. This can also be used to cross-check with/against app utilization metrics.
Rating of app | 3 months, 6 months
  Users are asked to rate the value of 8 different features of the app on a 5-point Likert scale from very poor to excellent. Plus, an overall rating of the likelihood of continued use of the app on a 5-point Likert scale from definitely not to definitely.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra E Moll, PhD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Western University, London, Ontario
  - Wilfrid Laurier University, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
May share aggregate utilisation data without personal identifiers.

REFERENCES:
- [Background] Zuromski KL, Ustun B, Hwang I, Keane TM, Marx BP, Stein MB, Ursano RJ, Kessler RC. Developing an optimal short-form of the PTSD Checklist for DSM-5 (PCL-5). Depress Anxiety. 2019 Sep;36(9):790-800. doi: 10.1002/da.22942. Epub 2019 Jul 29. PMID 31356709
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ramkissoon A, Smith P, Oudyk J. Dissecting the effect of workplace exposures on workers' rating of psychological health and safety. Am J Ind Med. 2019 May;62(5):412-421. doi: 10.1002/ajim.22964. Epub 2019 Mar 27. PMID 30916413
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Plouffe RA, Nazarov A, Forchuk CA, Gargala D, Deda E, Le T, Bourret-Gheysen J, Jackson B, Soares V, Hosseiny F, Smith P, Roth M, MacDougall AG, Marlborough M, Jetly R, Heber A, Albuquerque J, Lanius R, Balderson K, Dupuis G, Mehta V, Richardson JD. Impacts of morally distressing experiences on the mental health of Canadian health care workers during the COVID-19 pandemic. Eur J Psychotraumatol. 2021 Nov 10;12(1):1984667. doi: 10.1080/20008198.2021.1984667. eCollection 2021. PMID 34777712
- [Background] Pavolini E, Kuhlmann E, Agartan TI, Burau V, Mannion R, Speed E. Healthcare governance, professions and populism: Is there a relationship? An explorative comparison of five European countries. Health Policy. 2018 Oct;122(10):1140-1148. doi: 10.1016/j.healthpol.2018.08.020. Epub 2018 Sep 7. PMID 30219372
- [Background] Norman M, Ricciardelli R. Operational and organisational stressors in community correctional work: Insights from probation and parole officers in Ontario, Canada. Probat J. 2022 Mar;69(1):86-106. doi: 10.1177/0264550520984253. Epub 2021 Feb 3. PMID 35340787
- [Background] Moll SE, Patten S, Stuart H, MacDermid JC, Kirsh B. Beyond Silence: A Randomized, Parallel-Group Trial Exploring the Impact of Workplace Mental Health Literacy Training with Healthcare Employees. Can J Psychiatry. 2018 Dec;63(12):826-833. doi: 10.1177/0706743718766051. Epub 2018 Apr 19. PMID 29673271
- [Background] Moll S, Zanhour M, Patten SB, Stuart H, MacDermid J. Evaluating Mental Health Literacy in the Workplace: Development and Psychometric Properties of a Vignette-Based Tool. J Occup Rehabil. 2017 Dec;27(4):601-611. doi: 10.1007/s10926-017-9695-0. PMID 28120136
- [Background] Levis B, Sun Y, He C, Wu Y, Krishnan A, Bhandari PM, Neupane D, Imran M, Brehaut E, Negeri Z, Fischer FH, Benedetti A, Thombs BD; Depression Screening Data (DEPRESSD) PHQ Collaboration; Che L, Levis A, Riehm K, Saadat N, Azar M, Rice D, Boruff J, Kloda L, Cuijpers P, Gilbody S, Ioannidis J, McMillan D, Patten S, Shrier I, Ziegelstein R, Moore A, Akena D, Amtmann D, Arroll B, Ayalon L, Baradaran H, Beraldi A, Bernstein C, Bhana A, Bombardier C, Buji RI, Butterworth P, Carter G, Chagas M, Chan J, Chan LF, Chibanda D, Cholera R, Clover K, Conway A, Conwell Y, Daray F, de Man-van Ginkel J, Delgadillo J, Diez-Quevedo C, Fann J, Field S, Fisher J, Fung D, Garman E, Gelaye B, Gholizadeh L, Gibson L, Goodyear-Smith F, Green E, Greeno C, Hall B, Hampel P, Hantsoo L, Haroz E, Harter M, Hegerl U, Hides L, Hobfoll S, Honikman S, Hudson M, Hyphantis T, Inagaki M, Ismail K, Jeon HJ, Jette N, Khamseh M, Kiely K, Kohler S, Kohrt B, Kwan Y, Lamers F, Asuncion Lara M, Levin-Aspenson H, Lino V, Liu SI, Lotrakul M, Loureiro S, Lowe B, Luitel N, Lund C, Marrie RA, Marsh L, Marx B, McGuire A, Mohd Sidik S, Munhoz T, Muramatsu K, Nakku J, Navarrete L, Osorio F, Patel V, Pence B, Persoons P, Petersen I, Picardi A, Pugh S, Quinn T, Rancans E, Rathod S, Reuter K, Roch S, Rooney A, Rowe H, Santos I, Schram M, Shaaban J, Shinn E, Sidebottom A, Simning A, Spangenberg L, Stafford L, Sung S, Suzuki K, Swartz R, Tan PLL, Taylor-Rowan M, Tran T, Turner A, van der Feltz-Cornelis C, van Heyningen T, van Weert H, Wagner L, Li Wang J, White J, Winkley K, Wynter K, Yamada M, Zhi Zeng Q, Zhang Y. Accuracy of the PHQ-2 Alone and in Combination With the PHQ-9 for Screening to Detect Major Depression: Systematic Review and Meta-analysis. JAMA. 2020 Jun 9;323(22):2290-2300. doi: 10.1001/jama.2020.6504. PMID 32515813
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] King DK, Shoup JA, Raebel MA, Anderson CB, Wagner NM, Ritzwoller DP, Bender BG. Planning for Implementation Success Using RE-AIM and CFIR Frameworks: A Qualitative Study. Front Public Health. 2020 Mar 3;8:59. doi: 10.3389/fpubh.2020.00059. eCollection 2020. PMID 32195217
- [Background] Keith RE, Crosson JC, O'Malley AS, Cromp D, Taylor EF. Using the Consolidated Framework for Implementation Research (CFIR) to produce actionable findings: a rapid-cycle evaluation approach to improving implementation. Implement Sci. 2017 Feb 10;12(1):15. doi: 10.1186/s13012-017-0550-7. PMID 28187747
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Heber A, Testa V, Smith-MacDonald L, Bremault-Phillips S, Smith-MacDonald L. Rapid response to COVID-19: addressing challenges and increasing the mental readiness of public safety personnel. Health Promot Chronic Dis Prev Can. 2020 Dec 9;40(11-12):350-355. doi: 10.24095/hpcdp.40.11/12.04. Epub 2020 Sep 9. PMID 32909935
- [Background] Greenhalgh T, Wherton J, Papoutsi C, Lynch J, Hughes G, A'Court C, Hinder S, Fahy N, Procter R, Shaw S. Beyond Adoption: A New Framework for Theorizing and Evaluating Nonadoption, Abandonment, and Challenges to the Scale-Up, Spread, and Sustainability of Health and Care Technologies. J Med Internet Res. 2017 Nov 1;19(11):e367. doi: 10.2196/jmir.8775. PMID 29092808
- [Background] De Vito Dabbs A, Myers BA, Mc Curry KR, Dunbar-Jacob J, Hawkins RP, Begey A, Dew MA. User-centered design and interactive health technologies for patients. Comput Inform Nurs. 2009 May-Jun;27(3):175-83. doi: 10.1097/NCN.0b013e31819f7c7c. PMID 19411947
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Carleton RN, Afifi TO, Turner S, Taillieu T, Duranceau S, LeBouthillier DM, Sareen J, Ricciardelli R, MacPhee RS, Groll D, Hozempa K, Brunet A, Weekes JR, Griffiths CT, Abrams KJ, Jones NA, Beshai S, Cramm HA, Dobson KS, Hatcher S, Keane TM, Stewart SH, Asmundson GJG. Mental Disorder Symptoms among Public Safety Personnel in Canada. Can J Psychiatry. 2018 Jan;63(1):54-64. doi: 10.1177/0706743717723825. Epub 2017 Aug 28. PMID 28845686
- [Background] Carleton RN, Afifi TO, Taillieu T, Turner S, Mason JE, Ricciardelli R, McCreary DR, Vaughan AD, Anderson GS, Krakauer RL, Donnelly EA, Camp RD 2nd, Groll D, Cramm HA, MacPhee RS, Griffiths CT. Assessing the Relative Impact of Diverse Stressors among Public Safety Personnel. Int J Environ Res Public Health. 2020 Feb 14;17(4):1234. doi: 10.3390/ijerph17041234. PMID 32075062
- [Background] Anderson GS, Di Nota PM, Groll D, Carleton RN. Peer Support and Crisis-Focused Psychological Interventions Designed to Mitigate Post-Traumatic Stress Injuries among Public Safety and Frontline Healthcare Personnel: A Systematic Review. Int J Environ Res Public Health. 2020 Oct 20;17(20):7645. doi: 10.3390/ijerph17207645. PMID 33092146
- [Background] Richardson, J. D., Darte, K., Grenier, S., English, A., & Sharpe, J. (2008). Operational stress injury social support: A Canadian innovation in professional peer support. Canadian Military Journal, 9, 57-64.
- [Background] Ricciardelli, R., Groll, D., Czarnuch, S., Carleton, R. N., & Cramm, H. . (2019). Behind the frontlines: Exploring the mental health and help-seeking behaviours of public safety personnel who work to support frontline operations. Annual Review of Interdisciplinary Justice Research, 8, 315-348.
- [Background] Ricciardelli, R., Carleton, R. N., Cramm, H., & Groll, D. (2018). Qualitatively Unpacking Canadian Public Safety Personnel Experiences of Trauma and their Wellbeing: Physical Manifestations, Psychological Implications, and Fatalistic Attitudes. Canadian Journal of Criminology and Criminal Justice, 60, 566-577. Doi: 10.3138/cjccj.2017-0053.r2
- [Background] Ricciardelli, R. (2022). Informing Correctional Officer Discretion: A Co-Response Model and the Legal Vulnerabilities Inherent in Prison Work. The Prison Journal, 102(6), 651-672.
- [Background] Mehdizadeh, S., & Kamkar, K. (2020). COVID-19 and the impact on police services. Journal of Community Safety & Well-Being, 5, 42-44. Doi: 10.35502/jcswb.139
- [Background] Chalmers, L., & Keown, P. (2006). Communities of practice and professional development. International Journal of Lifelong Education, 25(2), 139-156. Doi: 10.1080/02601370500510793
- [Background] Carleton RN, Afifi TO, Turner S, Taillieu T, Vaughan AD, Anderson GS, Ricciardelli R, MacPhee RS, Cramm HA, Czarnuch S, Hozempa K, Camp RD. Mental health training, attitudes toward support, and screening positive for mental disorders. Cogn Behav Ther. 2020 Jan;49(1):55-73. doi: 10.1080/16506073.2019.1575900. Epub 2019 Feb 22. PMID 30794073
- [Background] Carleton, R. N., Afifi, T.O., Turner, S., Taillieu, T., LeBouthiller, D.M., Duranceau, S., Sareen, J., Ricciardelli, R., MacPhee, Krakauer, R., Anderson, G. S., Cramm, H. A., Groll, D., & McCreary, D. R. (2019). Exposures to potentially traumatic events among public safety personnel in Canada. Canadian Journal of Behavioural Science / Revue canadienne des sciences du comportement, 51(1), 37-52. Doi: 10.1037/cbs0000115
- [Background] Ricciardelli, R., Bucerius, S., Tetrault, J., Crewe, B., & Pyrooz, D. (2021). Correctional services during and beyond COVID-19. FACETS. 6. 490-516. Doi: 10.1139/facets-2021-0023.
- [Background] Oliphant, R. (2016). Healthy Minds, Safe Communities. Supporting Our Public Safety Officers Through a National Strategy for Operational Stress Injuries. Report of the Standing Committee on Public Safety and National Security. Ottawa, ON: House of Commons.
- [Background] American Psychiatric Association. (2013). Diagnostic and Statistical Manual of Mental Disorders (5th ed.). Washington, DC: Author.
- [Background] Canadian Institute for Public Safety Research and Treatment (CIPSRT). (2019). Glossary of terms: A shared understanding of the common terms used to describe psychological trauma (version 2.0). Regina, SK: Author.
- See also: Estimated Veteran Population by Province — https://www.veterans.gc.ca/eng/about-vac/news-media/facts-figures/1-0
- See also: CIPSRT COVID-19 Readiness Resource Project (CRRP) — https://www.cipsrt-icrtsp.ca/en/crrp